CLINICAL TRIAL: NCT00812981
Title: Non-inferiority Study of GSK Biologicals' Pandemic Influenza Vaccine 1562902A.
Brief Title: A Study for Evaluation of GSK Biologicals' Pandemic Influenza Vaccine.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 111954
Record Dates: First submitted 2008-12-18; First posted 2008-12-22 (Estimated); Results first posted 2017-06-16 (Actual); Last update posted 2018-08-20 (Actual); Status verified 2017-03

CONDITIONS: Influenza
Keywords: Pandemic influenza
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (2):
- 1562902A NP GROUP (Experimental): Healthy male or female adults, between and including 18 to 60 years of age, who received two doses of the new-processed (NP) 1562902A vaccine, administered intramuscularly in the deltoid region of the non-dominant arm, at Days 0 and 21.
  Interventions: Biological: GSK1562902A
- 1562902A CP GROUP (Experimental): Healthy male or female adults, between and including 18 to 60 years of age, who received two doses of the comparative-processed (CP) 1562902A vaccine, administered intramuscularly in the deltoid region of the non-dominant arm, at Days 0 and 21.
  Interventions: Biological: GSK1562902A

INTERVENTIONS:
Biological: GSK1562902A — new-processed (NP), administered intramuscularly in the deltoid region of the non-dominant arm
  Arms: 1562902A NP GROUP
Biological: GSK1562902A — comparative-processed (CP), administered intramuscularly in the deltoid region of the non-dominant arm
  Arms: 1562902A CP GROUP

SUMMARY:
This observer-blind study is designed to show the immunological non-inferiority of Thiomersal-free-processed pandemic influenza vaccine as compared to the Thiomersal-containing-processed pandemic influenza vaccine.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes that they can and will comply with the requirements of the protocol should be enrolled in the study.
* A male or female aged 18 to 60 years at the time of the first vaccination.
* Written informed consent obtained from the subject.
* Good general health as established by medical history and clinical examination before entering into the study.
* Access to a consistent means of telephone contact, which may be either in the home or at the workplace, land line or mobile, but NOT a pay phone or other multiple-user device
* Comprehension of the study requirements, ability to comprehend and comply with procedures for collection of short- and long-term safety data, expressed availability for the required study period, and ability and willingness to attend scheduled visits.
* If the subject is female, she must be of non-childbearing potential, or if she is of childbearing potential, she must practice adequate contraception for 30 days prior to vaccination, have a negative pregnancy test and continue such precautions for 2 months after completion of the vaccination series.

Exclusion Criteria:

* Evidence of substance abuse or of neurological or psychiatric diagnoses which, even if clinically stable, are deemed by the investigator to render the potential subject unable/unlikely to provide accurate safety reports.
* Diagnosed with cancer, or treatment for cancer, within 3 years.
* An oral temperature ≥ 37.8 º C or acute symptoms greater than "mild" severity on the scheduled date of first vaccination.
* Any confirmed or suspected immunosuppressive or immunodeficient condition including history of human immunodeficiency virus (HIV) infection.
* Receipt of systemic glucocorticoids (prednisone ≥ 5 mg/kg/day for more than 14 consecutive days) within 1 month of study enrolment, or any other cytotoxic or immunosuppressive drug within 6 months of study enrolment.
* Any significant disorder of coagulation or treatment with Coumarin derivatives or Heparin.
* Administration of any vaccines within 30 days before study enrolment.
* Previous administration of any H5N1 vaccine.
* Previous administration of vaccines with adjuvants similar to those used in the investigational vaccine.
* Use of any investigational or non-registered product (drug or vaccine) or planned participation in another investigational study within 30 days prior to study enrolment, or during the 180 days following the first test article dose. Use of any investigational or non-registered product with immunosuppressive properties is exclusionary at any time during the trial.
* Receipt of any immunoglobulins and/or any blood products within 3 months of study enrolment or planned administration of any of these products during the study period.
* Any known or suspected allergy to any constituent of influenza vaccines (including egg proteins or mercurial preservatives); a history of anaphylactic-type reaction to consumption of eggs; or a history of severe adverse reaction to a previous influenza vaccine.
* Known pregnancy or a positive urine beta-human chorionic gonadotropin (β-hCG) test result prior to either vaccination.
* Lactating women.
* Women of child bearing potential who lack a history of reliable contraceptive practices. The provision of this history does NOT replace the requirement to perform, and obtain negative results in pregnancy urine tests prior to treatments.
* Known use of an analgesic or antipyretic medication within 12 hours prior to first treatment.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 320 (Actual)
Dates: Start 2008-11-15 (Actual); Primary Completion 2009-06-07 (Actual); Study Completion 2009-06-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Yang PC, Yu CJ, Chang SC, Hsieh SM, Drame M, Walravens K, Roman F, Gillard P. Safety and immunogenicity of a split-virion AS03A-adjuvanted A/Indonesia/05/2005 (H5N1) vaccine in Taiwanese adults. J Formos Med Assoc. 2012 Jun;111(6):333-9. doi: 10.1016/j.jfma.2011.02.006. Epub 2012 Apr 20. PMID 22748624
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Study Protocol: 111954 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 111954 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 111954 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 111954 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 111954 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 111954 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 111954 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 1562902A NP Group | 1562902A CP Group
Started | 160 | 160
Completed | 160 | 159
Not Completed | 0 | 1
Not completed — Other | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1562902A NP Group | 1562902A CP Group | Total
Number analyzed (Participants) | 160 | 160 | 320
Age, Continuous [Mean (Standard Deviation); unit: Years] | 31.30 (7.95) | 32.60 (9.10) | 31.95 (8.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 80 | 83 | 163
  Male | 80 | 77 | 157
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian - East-Asian heritage | 160 | 160 | 320

OUTCOME MEASURES:

1. Primary Outcome: Titers for Serum H5N1 Haemagglutination-inhibition (HI) Antibodies
Description: Titers are presented as geometric mean titers (GMTs). The reference seropositivity cut-off value was equal to or above (≥) 1:10. The flu strain assessed was A/Indonesia/05/2005.
Time Frame: At Day 42
Population: The analysis was performed on the ATP cohort for immunogenicity, which included all evaluable subjects for whom data concerning immunogenicity outcome variables were available.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | 1562902A NP Group | 1562902A CP Group
Number analyzed (Participants) | 156 | 155
Titers | 739.5 [667.8 to 818.8] | 621.7 [542.9 to 712.0]
Statistical Analysis 1: Comparison: 1562902A NP Group vs 1562902A CP Group; Difference in adjusted GMT ratio for HI antibodies: To demonstrate that the NP 1562902A vaccine was non-inferior to the CP 1562902A vaccine, with respect to HI antibody GMT against the A/Indonesia/05/2005 strain, 42 days following vaccination; Test type: Non-Inferiority or Equivalence — Non-inferiority was defined as the upper limit of the two-sided 95% confidence interval (CI) for the GMT ratio of HI antibodies against the A/Indonesia/05/2005 strain between the two groups (1562902A CP Group over 1562902A NP Group), being below (<) 2.0; ANCOVA; Adjusted GMT ratio = 0.84, 95% CI 2-sided [0.71 to 0.99]

2. Secondary Outcome: Titers for Serum H5N1 HI Antibodies
Description: Titers are presented as geometric mean titers (GMTs). The reference seropositivity cut-off value was equal to or above (≥) 1:10. The flu strains assessed were A/Indonesia/05/2005 and A/Vietnam/1194/2004.
Time Frame: At Day 0 and Day 180
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | 1562902A NP Group | 1562902A CP Group
Number analyzed (Participants) | 156 | 156
Titers
  A/Indonesia/05/2005, Day 0 | 5.0 [5.0 to 5.0] | 5.1 [5.0 to 5.2]
  A/Indonesia/05/2005, Day 180: number analyzed (Participants) | 156 | 155
  A/Indonesia/05/2005, Day 180 | 51.9 [45.1 to 59.7] | 33.0 [28.0 to 39.0]
  A/Vietnam/1194/2004, Day 0 | 5.1 [4.9 to 5.3] | 5.2 [5.0 to 5.5]
  A/Vietnam/1194/2004, Day 180: number analyzed (Participants) | 156 | 155
  A/Vietnam/1194/2004, Day 180 | 12.6 [10.8 to 14.8] | 8.4 [7.3 to 9.5]

3. Secondary Outcome: Number of Subjects With H5N1 HI Antibody Concentrations Above the Cut-off Value
Description: The cut-off values for the humoral immune response in terms of H5N1 HI antibodies were equal to or above (≥) 1:10. The flu strains assessed were A/Indonesia/05/2005 and A/Vietnam/1194/2004.
Time Frame: At Days 0, 42 and 180
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | 1562902A NP Group | 1562902A CP Group
Number analyzed (Participants) | 156 | 156
Participants
  A/Indonesia/05/2005, Day 0 | 0 | 3
  A/Indonesia/05/2005, Day 42: number analyzed (Participants) | 156 | 155
  A/Indonesia/05/2005, Day 42 | 156 | 154
  A/Indonesia/05/2005, Day 180: number analyzed (Participants) | 156 | 155
  A/Indonesia/05/2005, Day 180 | 145 | 128
  A/Vietnam/1194/2004, Day 0 | 2 | 3
  A/Vietnam/1194/2004, Day 42: number analyzed (Participants) | 156 | 155
  A/Vietnam/1194/2004, Day 42 | 149 | 140
  A/Vietnam/1194/2004, Day 180: number analyzed (Participants) | 156 | 155
  A/Vietnam/1194/2004, Day 180 | 82 | 50

4. Secondary Outcome: Number of Seroconverted Subjects Against Two Strains of Influenza Disease
Description: A seroconverted subject was defined as a vaccinated subject who had either a pre-vaccination titer below (<) 1:10 and a post-vaccination titer equal to or above (≥) 1:40, or a pre-vaccination titer ≥ 1:10 and at least a four-fold increase in post-vaccination titer. The flu strains assessed were A/Indonesia/05/2005 and A/Vietnam/1194/2004.
Time Frame: At Day 42 and Day 180
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | 1562902A NP Group | 1562902A CP Group
Number analyzed (Participants) | 156 | 155
Participants
  A/Indonesia/05/2005, Day 42 | 156 | 153
  A/Indonesia/05/2005, Day 180 | 129 | 104
  A/Vietnam/1194/2004, Day 42 | 143 | 126
  A/Vietnam/1194/2004, Day 180 | 34 | 13

5. Secondary Outcome: Seroconversion Factor (SCF) for H5N1 HI Antibodies
Description: The seroconversion factor (SCF) was defined as the fold increase in H5N1 HI antibody GMTs post-vaccination compared to Day 0. The flu strains assessed were A/Indonesia/05/2005 and A/Vietnam/1194/2004.
Time Frame: At Day 42 and Day 180
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Fold change
Arm/Group | 1562902A NP Group | 1562902A CP Group
Number analyzed (Participants) | 156 | 155
Fold change
  A/Indonesia/05/2005, Day 42 | 147.9 [133.6 to 163.8] | 121.9 [106.3 to 139.7]
  A/Indonesia/05/2005, Day 180 | 10.4 [9.0 to 11.9] | 6.5 [5.5 to 7.6]
  A/Vietnam/1194/2004, Day 42 | 15.6 [13.5 to 17.9] | 10.8 [9.1 to 12.7]
  A/Vietnam/1194/2004, Day 180 | 2.5 [2.1 to 2.9] | 1.6 [1.4 to 1.8]

6. Secondary Outcome: Number of Seroprotected Subjects for H5N1 HI Antibodies
Description: A seroprotected subject was defined as a vaccinated subject with a serum HI titer equal to or above (≥) 1:40. The flu strains assessed were A/Indonesia/05/2005 and A/Vietnam/1194/2004.
Time Frame: At Days 0, 42 and 180
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | 1562902A NP Group | 1562902A CP Group
Number analyzed (Participants) | 156 | 156
Participants
  A/Indonesia/05/2005, Day 0 | 0 | 0
  A/Indonesia/05/2005, Day 42 | 156 | 153
  A/Indonesia/05/2005, Day 180 | 129 | 104
  A/Vietnam/1194/2004, Day 0 | 1 | 3
  A/Vietnam/1194/2004, Day 42 | 144 | 127
  A/Vietnam/1194/2004, Day 180 | 34 | 16

7. Secondary Outcome: Titers for Serum Neutralising Antibodies Against A/Vietnam/1194/2004 Strain of Influenza Disease
Description: Titers are presented as geometric mean titers (GMTs). The reference seropositivity cut-off value was equal to or above (≥) 1:28. The flu strain assessed was A/Vietnam/1194/2004.
Time Frame: At Days 0, 42 and 180
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | 1562902A NP Group | 1562902A CP Group
Number analyzed (Participants) | 58 | 60
Titers
  A/Vietnam/1194/2004, Day 0 | 189.1 [149.8 to 238.7] | 166.3 [135.4 to 204.2]
  A/Vietnam/1194/2004, Day 42: number analyzed (Participants) | 58 | 59
  A/Vietnam/1194/2004, Day 42 | 376.7 [308.2 to 460.4] | 359.2 [320.9 to 402.0]
  A/Vietnam/1194/2004, Day 180: number analyzed (Participants) | 58 | 59
  A/Vietnam/1194/2004, Day 180 | 184.5 [151.6 to 224.6] | 197.3 [159.6 to 244.0]

8. Secondary Outcome: Number of Subjects With Neutralizing Antibody Concentrations Above the Cut-off Value
Description: Seropositivity cut-off values assessed were equal to or above (≥) 1:28 in the sera of subjects seronegative before vaccination. The flu strain assessed was A/Vietnam/1194/2004.
Time Frame: At Days 0, 42 and 180
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | 1562902A NP Group | 1562902A CP Group
Number analyzed (Participants) | 58 | 60
Participants
  A/Vietnam/1194/2004, Day 0 | 56 | 59
  A/Vietnam/1194/2004, Day 42: number analyzed (Participants) | 58 | 59
  A/Vietnam/1194/2004, Day 42 | 57 | 59
  A/Vietnam/1194/2004, Day 180: number analyzed (Participants) | 58 | 59
  A/Vietnam/1194/2004, Day 180 | 57 | 59

9. Secondary Outcome: Number of Seroconverted Subjects for Neutralizing Antibodies
Description: A seroconverted subject was defined as a vaccinated subject who had either a pre-vaccination titer < 1:28 and a post-vaccination titer ≥ 1:56 or a pre-vaccination titer ≥ 1:28 and at least a four-fold increase in post-vaccination titer. The flu strain assessed was A/Vietnam/1194/2004.
Time Frame: At Day 42 and Day 180
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | 1562902A NP Group | 1562902A CP Group
Number analyzed (Participants) | 58 | 59
Participants
  A/Vietnam/1194/2004, Day 42 | 15 | 13
  A/Vietnam/1194/2004, Day 180 | 7 | 9

10. Secondary Outcome: Number of Subjects With Any and Grade 3 Solicited Local Symptoms
Description: Assessed solicited local symptoms were pain, redness and swelling. Any = occurrence of the symptom regardless of intensity grade. Grade 3 pain = pain that prevented normal activity. Grade 3 redness/swelling = redness/swelling spreading beyond 100 millimeters (mm) of injection site.
Time Frame: During the 7-day (Days 0-6) post-vaccination period following each dose and across doses
Population: The analysis was performed on the Total Vaccinated Cohort, which included all vaccinated subjects for whom safety data were available and who had the symptom sheet filled in.
Measure: Count of Participants; unit: Participants
Arm/Group | 1562902A NP Group | 1562902A CP Group
Number analyzed (Participants) | 160 | 159
Participants
  Any Pain, Dose 1 | 141 | 137
  Grade 3 Pain, Dose 1 | 9 | 4
  Any Redness, Dose 1 | 3 | 2
  Grade 3 Redness, Dose 1 | 0 | 0
  Any Swelling, Dose 1 | 13 | 14
  Grade 3 Swelling, Dose 1 | 0 | 0
  Any Pain, Dose 2: number analyzed (Participants) | 159 | 157
  Any Pain, Dose 2 | 137 | 133
  Grade 3 Pain, Dose 2: number analyzed (Participants) | 159 | 157
  Grade 3 Pain, Dose 2 | 9 | 4
  Any Redness, Dose 2: number analyzed (Participants) | 159 | 157
  Any Redness, Dose 2 | 4 | 3
  Grade 3 Redness, Dose 2: number analyzed (Participants) | 159 | 157
  Grade 3 Redness, Dose 2 | 0 | 0
  Any Swelling, Dose 2: number analyzed (Participants) | 159 | 157
  Any Swelling, Dose 2 | 17 | 12
  Grade 3 Swelling, Dose 2: number analyzed (Participants) | 159 | 157
  Grade 3 Swelling, Dose 2 | 0 | 2
  Any Pain, Across doses | 152 | 146
  Grade 3 Pain, Across doses | 12 | 8
  Any Redness, Across doses | 4 | 5
  Grade 3 Redness, Across doses | 0 | 0
  Any Swelling, Across doses | 21 | 19
  Grade 3 Swelling, Across doses | 0 | 2

11. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Solicited General Symptoms
Description: Assessed solicited general symptoms were arthralgia, fatigue, headache, myalgia, shivering, sweating and fever [defined as axillary temperature equal to or above (≥) 38 degrees Celsius (°C)]. Any = occurrence of the symptom regardless of intensity grade. Grade 3 symptom = symptom that prevented normal activity. Grade 3 fever = fever ≥ 39.0 °C. Related = symptom assessed by the investigator as causally related to the study vaccination.
Time Frame: During the 7-day (Days 0-6) post-vaccination period following each dose and across doses
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | 1562902A NP Group | 1562902A CP Group
Number analyzed (Participants) | 160 | 159
Participants
  Any Arthralgia, Dose 1 | 10 | 14
  Grade 3 Arthralgia, Dose 1 | 0 | 0
  Related Arthralgia, Dose 1 | 10 | 13
  Any Fatigue, Dose 1 | 62 | 68
  Grade 3 Fatigue, Dose 1 | 2 | 2
  Related Fatigue, Dose 1 | 60 | 65
  Any Headache, Dose 1 | 31 | 43
  Grade 3 Headache, Dose 1 | 1 | 2
  Related Headache, Dose 1 | 27 | 40
  Any Myalgia, Dose 1 | 90 | 78
  Grade 3 Myalgia, Dose 1 | 2 | 2
  Related Myalgia, Dose 1 | 88 | 75
  Any Shivering, Dose 1 | 2 | 4
  Grade 3 Shivering, Dose 1 | 0 | 0
  Related Shivering, Dose 1 | 2 | 4
  Any Sweating, Dose 1 | 9 | 10
  Grade 3 Sweating, Dose 1 | 0 | 0
  Related Sweating, Dose 1 | 9 | 8
  Any Fever, Dose 1 | 0 | 4
  Grade 3 Fever, Dose 1 | 0 | 1
  Related Fever, Dose 1 | 0 | 4
  Any Arthralgia, Dose 2: number analyzed (Participants) | 159 | 157
  Any Arthralgia, Dose 2 | 27 | 27
  Grade 3 Arthralgia, Dose 2: number analyzed (Participants) | 159 | 157
  Grade 3 Arthralgia, Dose 2 | 2 | 2
  Related Arthralgia, Dose 2: number analyzed (Participants) | 159 | 157
  Related Arthralgia, Dose 2 | 26 | 27
  Any Fatigue, Dose 2: number analyzed (Participants) | 159 | 157
  Any Fatigue, Dose 2 | 87 | 82
  Grade 3 Fatigue, Dose 2: number analyzed (Participants) | 159 | 157
  Grade 3 Fatigue, Dose 2 | 8 | 4
  Related Fatigue, Dose 2: number analyzed (Participants) | 159 | 157
  Related Fatigue, Dose 2 | 87 | 82
  Any Headache, Dose 2: number analyzed (Participants) | 159 | 157
  Any Headache, Dose 2 | 51 | 49
  Grade 3 Headache, Dose 2: number analyzed (Participants) | 159 | 157
  Grade 3 Headache, Dose 2 | 4 | 2
  Related Headache, Dose 2: number analyzed (Participants) | 159 | 157
  Related Headache, Dose 2 | 51 | 49
  Any Myalgia, Dose 2: number analyzed (Participants) | 159 | 157
  Any Myalgia, Dose 2 | 67 | 62
  Grade 3 Myalgia, Dose 2: number analyzed (Participants) | 159 | 157
  Grade 3 Myalgia, Dose 2 | 7 | 3
  Related Myalgia, Dose 2: number analyzed (Participants) | 159 | 157
  Related Myalgia, Dose 2 | 66 | 62
  Any Shivering, Dose 2: number analyzed (Participants) | 159 | 157
  Any Shivering, Dose 2 | 16 | 11
  Grade 3 Shivering, Dose 2: number analyzed (Participants) | 159 | 157
  Grade 3 Shivering, Dose 2 | 2 | 0
  Related Shivering, Dose 2: number analyzed (Participants) | 159 | 157
  Related Shivering, Dose 2 | 16 | 11
  Any Sweating, Dose 2: number analyzed (Participants) | 159 | 157
  Any Sweating, Dose 2 | 11 | 11
  Grade 3 Sweating, Dose 2: number analyzed (Participants) | 159 | 157
  Grade 3 Sweating, Dose 2 | 0 | 0
  Related Sweating, Dose 2: number analyzed (Participants) | 159 | 157
  Related Sweating, Dose 2 | 11 | 10
  Any Fever, Dose 2: number analyzed (Participants) | 159 | 157
  Any Fever, Dose 2 | 10 | 12
  Grade 3 Fever, Dose 2: number analyzed (Participants) | 159 | 157
  Grade 3 Fever, Dose 2 | 1 | 1
  Related Fever, Dose 2: number analyzed (Participants) | 159 | 157
  Related Fever, Dose 2 | 10 | 12
  Any Arthralgia, Across doses | 32 | 33
  Grade 3 Arthralgia, Across doses | 2 | 2
  Related Arthralgia, Across doses | 31 | 32
  Any Fatigue, Across doses | 104 | 99
  Grade 3 Fatigue, Across doses | 9 | 6
  Related Fatigue, Across doses | 102 | 98
  Any Headache, Across doses | 59 | 68
  Grade 3 Headache, Across doses | 4 | 4
  Related Headache, Across doses | 59 | 67
  Any Myalgia, Across doses | 110 | 101
  Grade 3 Myalgia, Across doses | 8 | 5
  Related Myalgia, Across doses | 109 | 101
  Any Shivering, Across doses | 16 | 14
  Grade 3 Shivering, Across doses | 2 | 0
  Related Shivering, Across doses | 16 | 14
  Any Sweating, Across doses | 16 | 18
  Grade 3 Sweating, Across doses | 0 | 0
  Related Sweating, Across doses | 16 | 15
  Any Fever, Across doses | 10 | 16
  Grade 3 Fever, Across doses | 1 | 2
  Related Fever, Across doses | 10 | 16

12. Secondary Outcome: Number of Subjects With Any Adverse Events of Specific Interest (AESIs)
Description: An AESI was defined as an AE including autoimmune diseases and other mediated inflammatory disorders and assessed by the investigator as specific to the treatment administration.
Time Frame: From Day 0 up to 51 days after the first vaccination
Population: The analysis was performed on the Total Vaccinated Cohort which included all vaccinated subjects for whom safety data were available.
Measure: Count of Participants; unit: Participants
Arm/Group | 1562902A NP Group | 1562902A CP Group
Number analyzed (Participants) | 160 | 160
Participants | 1 | 0

13. Secondary Outcome: Number of Subjects With Any AESIs
Description: as for outcome 12
Time Frame: During the entire study period (from Day 0 up to Day 180)
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | 1562902A NP Group | 1562902A CP Group
Number analyzed (Participants) | 160 | 160
Participants | 1 | 0

14. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Unsolicited Adverse Events (AEs)
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination. Grade 3 AE = an AE which prevented normal, everyday activities. Related = AE assessed by the investigator as related to the vaccination.
Time Frame: During the 21-day follow-up period after the first vaccination and 30-day follow-up period after the second vaccination
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | 1562902A NP Group | 1562902A CP Group
Number analyzed (Participants) | 160 | 160
Participants
  Any AE(s) | 49 | 53
  Grade 3 AE(s) | 4 | 8
  Related AE(s) | 15 | 12

15. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Unsolicited Adverse Events (AEs)
Description: as for outcome 14
Time Frame: During the entire study period (from Day 0 up to Day 180)
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | 1562902A NP Group | 1562902A CP Group
Number analyzed (Participants) | 160 | 160
Participants
  Any AE(s) | 54 | 62
  Grade 3 AE(s) | 5 | 8
  Related AE(s) | 15 | 12

16. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: SAEs assessed include medical occurrences that result in death, are life-threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity.
Time Frame: From Day 0 up to Day 51
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | 1562902A NP Group | 1562902A CP Group
Number analyzed (Participants) | 160 | 160
Participants | 3 | 0

17. Secondary Outcome: Number of Subjects With SAEs
Description: as for outcome 16
Time Frame: During the entire study period (from Day 0 up to Day 180)
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | 1562902A NP Group | 1562902A CP Group
Number analyzed (Participants) | 160 | 160
Participants | 4 | 2

ADVERSE EVENTS:
Time Frame: Solicited local and general symptoms: during the 7-day (Days 0-6) post-vaccination period; Unsolicited AEs and SAEs: during the entire study period (from Day 0 up to Day 180).
Arm/Group | 1562902A NP Group | 1562902A CP Group
All-Cause Mortality (participants affected / at risk) | 0/160 | 0/160
Serious Adverse Events (participants affected / at risk) | 4/160 | 2/160
Other Adverse Events (participants affected / at risk) | 155/160 | 150/160
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 1562902A NP Group (N=160) | 1562902A CP Group (N=160)
Calculus urinary (Renal and urinary disorders) | 1 | 0
Endometrial cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1
Injury (Injury, poisoning and procedural complications) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 1562902A NP Group (N=160) | 1562902A CP Group (N=160)
Pain (General disorders) | 152 | 146
Swelling (General disorders) | 21 | 19
Arthralgia (General disorders) | 32 | 33
Fatigue (General disorders) | 104 | 99
Headache (General disorders) | 59 | 68
Myalgia (General disorders) | 110 | 101
Shivering (General disorders) | 16 | 14
Sweating (General disorders) | 16 | 18
Fever (General disorders) | 10 | 16
Nasopharyngitis (Infections and infestations) | 20 | 27
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 9 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.